CLINICAL TRIAL: NCT06235450
Title: A Usability Study of iTEAR100 For Combined EyeLid Microblepharoexfoliation and Neurostimulation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olympic Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-012
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: MicroBlepharoexfoliation, NuLids, iTEAR100, iLIDS100, Blepharitis, Dry Eye Syndrome
MeSH Terms: conditions — Blepharitis; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Open Label, Prospective, Therapeutic Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic iLIDS arm (Experimental): Subjects apply iTEAR100 device with iLIDS100 accessory
  Interventions: Device: iLIDS100

INTERVENTIONS:
Device: iLIDS100 — Subject applies iLIDS accessory to the iTEAR100 device. Applies to Eyelid margin similar to commercial products

SUMMARY:
The purpose of this study is to evaluate the usability of the iTEAR100 generation 2 device in combination with its newly developed iLIDS100 disposable cover.

DETAILED DESCRIPTION:
This usability study is meant to validate treatment using the iLIDS100 in patients who already use the NuLids Device and iTEAR100. The patients will simply substitute the iLIDS100 cover in combination with the iTEAR100 for the NuLids product and otherwise maintain their same treatment regimen. The planned number of subjects was chosen to provide clinically relevant usability data

ELIGIBILITY:
Inclusion Criteria:

Must use iTEAR and NuLids at time of enrollment

Exclusion Criteria:

1. have any condition, which in the judgment of the PI would prevent a potential subject from safely completing the study or tolerating device use, such as mental illness, dementia, severe agitation, etc. and including inability to comply with the treatment regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 30 days
  How does iLids compare to NuLids product

CONTACTS AND LOCATIONS:
Locations (1):
- Olympic Ophthalmics, Issaquah, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Full dataset , 30 days after study close
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 30 days after study completion